CLINICAL TRIAL: NCT05728021
Title: Efficacy of a Therapist-guided Smartphone-based Intervention to Support Recovery From Bulimia Nervosa: a Randomized Controlled Multi-center Trial
Brief Title: Smartphone-based Aftercare for Inpatients With Bulimia Nervosa
Acronym: SMART-BN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Schoen Clinic Roseneck (Unknown); Schoen Clinic Bad Bramstedt (Unknown); Schoen Clinic Bad Arolsen (Unknown); Klinik Lüneburger Heide (Unknown); Else Kröner Fresenius Foundation (Other)
Responsible Party: Principal Investigator, Schlegl Sandra, Principal Investigator, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-084
Record Dates: First submitted 2020-09-09; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Bulimia Nervosa
Keywords: Bulimia nervosa; Smartphone; Aftercare; Inpatient
MeSH Terms: conditions — Bulimia Nervosa | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Record Aftercare (Experimental): Intervention group (IG)
  Interventions: Behavioral: Recovery Record Aftercare
- Treatment as usual (TAU) (Active Comparator): Control group (CG)
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Recovery Record Aftercare — Patients randomized to IG receive a therapist-guided smartphone-based aftercare intervention for a period of 16 weeks. The patients are invited to download for free the German version of "Recovery Record" at the App Store (iPhone) or the Google Play Store (android) to their smartphone and to link with the aftercare therapist. After discharge, patients are asked to monitor their meals at least three times per day (breakfast, lunch, and dinner), that is, to produce a minimum of three logs per day over the subsequent 16 weeks. Furthermore, patients are instructed to monitor their thoughts and feelings as well as their (eating disordered) behaviors. The aftercare therapist also sets the patients clinical post-discharge goals and makes coping skill suggestions. Individual therapist feedback is provided in-app twice per week during the first four weeks, once per week in weeks 5-8 and every other week in weeks 9-16.
  Arms: Recovery Record Aftercare
Behavioral: Treatment as usual (TAU) — Patients randomized to CG receive TAU i.e. patients and their physicians or therapists decide on post-discharge treatment which is documented at T1 and T2. Patients from the CG are also assessed at all assessment points.
  Arms: Treatment as usual (TAU)

SUMMARY:
Inpatient treatment for patients with bulimia nervosa (BN) is recommended in extreme or severe cases and/or after failure of outpatient treatment and is highly effective. However, a number of patients show symptom increase and relapse after discharge. The aim of this study is to evaluate the efficacy of a guided smartphone-based aftercare intervention following inpatient treatment of patients with BN to support recovery.

DETAILED DESCRIPTION:
Bulimia nervosa (BN) is a severe mental disorder characterized by recurrent episodes of binge eating and recurrent inappropriate compensatory behaviors to prevent weight gain. Evidence-based psychological treatments exist, however, even if treatment is successful in reducing behaviors such as binge eating and purging, abstinence rates may remain low and even if remission or abstinence have been received after treatment relapse rates are substantial. There is evidence that the stability of remission increases if the corresponding symptom improvement lasts at least for 4 months. Studies on the effectiveness of inpatient treatment in adult patients with BN show responder rates of up to 77%. However, it is often difficult for patients to maintain therapy success after discharge, as relapse rates reach up to 40% with the highest risk during the first 5 or 6 months after remission. There is preliminary evidence for efficacy regarding the potential of technology-based interventions in aftercare for patients with BN. However, so far, there is no study evaluating a smartphone-based aftercare intervention for patients with BN. Therefore, the aim of this study is to investigate the efficacy of a guided smartphone-based aftercare intervention as an add-on element to treatment as usual (TAU) compared to TAU alone in inpatients with BN. Our primary hypothesis is that the intervention group shows a significantly higher remission rate than TAU at end of treatment.

Eligible patients with BN who are discharged from inpatient treatment will be randomized either to receive a 4-month smartphone-based aftercare intervention with therapist feedback as an add-on element to treatment as usual (TAU) or TAU alone. Assessment points will be as follows: at hospital discharge (=baseline, T0), 16 weeks (=end of the aftercare intervention, T1) and after 10 months (=6-month follow-up, T2).

ELIGIBILITY:
Inclusion Criteria:

1. primary diagnosis of BN (DSM-5: 307.51) at admission as assessed by the diagnostically relevant items from the Eating Disorder Examination (Hilbert et al. 2016b),
2. sex: female,
3. age: from 13 years onwards to 60 years,
4. regular completion of inpatient treatment,
5. at least a length of inpatient stay of 6 weeks,
6. remission defined as less than once a week of binge eating and compensatory behavior in the past 28 days thus no longer meeting the full criteria for BN according to DSM-5,
7. owner of a smartphone,
8. informed consent of the patient and, in case of minors, also of the parents.

Exclusion Criteria:

1. major depression (Beck Depression Inventory-II (BDI-II) > 29 at discharge),
2. suicidal tendency (item 9 of BDI-II > 1 at discharge),
3. very high level of care after inpatient treatment (e.g. therapeutic living community, day clinic),
4. pregnancy.

Ages: 13 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Changes in Eating Disorder Severity (assessor-based) | Measured at baseline (discharge), at week 16 (end of treatment) and 6 month follow-up
  The Eating Disorder Examination (EDE) will be used to measure assessor-based eating disorder symptom severity over time. Minimum value: 0, maximum value: 6. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Changes in Eating Disorder Severity (self-report) | Measured at baseline, week 4, week 16 and 6 month follow-up
  The Eating Disorder Examination Questionnaire (EDE-Q) will be used to measure self-reported eating disorder symptom severity over time. Minimum value: 0, maximum value: 6. Higher scores mean a worse outcome.
Changes in Body-Mass-Index (BMI) | Measured at baseline, week 16 and 6 month follow-up
  Weight and height will be used to measure BMI over time.
Changes in depressive symptoms | Measured at baseline, week 16 and 6 month follow-up
  The Beck Depression Inventory-II (BDI-II) will be used to measure depressive symptoms. Minimal value: 0, maximum value: 63. Higher scores mean a worse outcome.
Changes in stages of change regarding specific eating disorder behaviors | Measured at baseline, week 16 and 6 month follow-up
  The Stages of Change Questionnaire for Eating Disorders (SOCQ-ED) will be used to measure changes in stages of change (precontemplation, contemplation, preparation, action, maintenance, termination) specific eating disorder behaviors over time.
Changes in general self-efficacy | Measured at baseline, week 16 and 6 month follow-up
  The General Self-Efficacy Scale (GSE) will be used to measure self-efficacy over time. Minimum value: 10, maximum value: 40. Higher scores mean a better outcome.
Changes in eating disorder specific self-efficacy | Measured at baseline, week 16 and 6 month follow-up
  A self-efficacy scale will be used to measure self-efficacy regarding patients' confidence about resisting binge eating over time. Minimum value: 0, maximum value: 3. Higher scores mean better outcomes.
Therapeutic Alliance | Measured at week 4 and week 16
  The Helping Alliance Questionnaire (HAQ) will be used to measure therapeutic alliance. Minimum value: 11, maximum value: 66. Higher scores mean a better outcome.
Ratings of suitability of treatment and expectancy of treatment outcome | Measured at week 4
  Ten-point visual analogue scales will assess patients' perceptions of the suitability of the aftercare intervention and their expectations that they would maintain their remission status. Higher scores mean a better suitability and expectancy.
Participant satisfaction with the app and the aftercare intervention | Measured at week 16
  A self-developed questionnaire will be used to assess self-reported satisfaction with the app and the aftercare intervention. Minimum value: 1, maximum value: 5. Higher scores mean a better satisfaction.
Additional outpatient and inpatient treatment after discharge | Measured at week 16 and 6 month follow-up
  Number and length of outpatient or inpatient treatment (rehospitalization) since discharge will be assessed.
Adherence to the smartphone-based aftercare intervention | Measured from baseline to week 16
  Adherence will be measured via dichotomous outcome of drop-out (individuals will be considered as drop-out if they fail to login to the app at all for a period of 14 consecutive days. Adherence will be assessed through application usage data.
Adherence to self-monitoring tasks | Measured from baseline to week 16
  Frequency of self-monitoring entries will be tracked automatically through the program server

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Schlegl, PhD, Principal Investigator — Ludwig Maximilian University Munich; Ulrich Voderholzer, MD, Principal Investigator — Schoen Clinic Roseneck
Locations (4):
- Germany (4):
  - Schoen Clinic Bad Arolsen, Bad Arolsen
  - Klinik Lüneburger Heide, Bad Bevensen
  - Schoen Clinic Bad Bramstedt, Bad Bramstedt
  - Schoen Clinic Roseneck, Prien am Chiemsee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ekfs.de/en/scientific-funding/currently-funded-projects/efficacy-therapist-guided-smartphone-based